CLINICAL TRIAL: NCT01602146
Title: Acute and Chronic Problems Associated With the Practice of Mountain Ultramarathon
Brief Title: Problems Associated With Ultramarathon
Acronym: CHAMONIX2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208048; 2012-A00424-39 (Other: AFSSAPS)
Record Dates: First submitted 2012-05-02; First posted 2012-05-18 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Ultramarathon Runner
Keywords: ultramarathon central fatigue,
MeSH Terms: interventions — Marathon Running

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultramarathon runner: People who do the Mont Blanc ultramarathon (31/08/12 to 02/09/12)
  Interventions: Other: ultramarathon running

INTERVENTIONS:
Other: ultramarathon running — * blood samples before and after ultramarathon
  * urinary samples before and after ultramarathon
  * voluntary ant electrically muscular forces measuring before and after ultramarathon
  * Broadband ultrasound Attenuation before and after ultramarathon

SUMMARY:
Acute physiological consequences of ultramarathon running are still unknown, particularly in women. Results from the investigators first studies conducted in 2009 have shown that a large part of fatigue induced by a mountain ultramarathon could be attributed to central fatigue. The investigators have investigated the biological consequences and neuromuscular fatigue only in male runners. Data from the literature suggest that amplitude and etiology of fatigue after prolonged exercise might be gender-dependant.The main purpose of the present project is thus to quantify supraspinal central fatigue and associated changes in cortical excitability after an extreme exercise such as a mountain ultramarathon: the Ultra-Trail du Mont-blanc, by using TMS.

DETAILED DESCRIPTION:
Acute physiological consequences of ultramarathon running are still unknown, particularly in women. Results from our first studies conducted in 2009 have shown that a large part of fatigue induced by a mountain ultramarathon could be attributed to central fatigue. Indeed, during extreme exercises such as 24h running, strength losses of knee extensor muscles have reached -40% and ¾ of this fatigue was explain by a central deficit while peripheral mechanisms explained only ¼. Similar results have been reported after a mountain ultramarathon despite the fact that several downhill have induced number of eccentric contractions. As a consequence, central fatigue must be particularly investigated. For this purpose, transcranial magnetic stimulation (TMS) has been recently validated to measure supraspinal central fatigue and cortical excitability.

We have investigated the biological consequences and neuromuscular fatigue only in male runners. Data from the literature suggest that amplitude and etiology of fatigue after prolonged exercise might be gender-dependant. However, these physiological data and studies that have paired male and female by level of performance on shorter distances seem contradictory with performance comparison between genders so that the relative superiority of women in ultra-endurance is not ascertained. The hypothesis of a greater fatigue resistance after ultramarathons in women should then be tested. The biological consequences of ultramarathon are far to be negligible in terms of inflammatory syndrome but complete characterization of this syndrome after such an extreme exercise has yet to be done. Also, several cases of renal failure have been reported after ultramarathons. Evaluation of ultramarathon consequences on kidneys is necessary to prevent serious complications. Finally, consequences of an ultramarathon are not only linked to races but also to training, i.e. the prolonged time spent in running to prepare for the races. Energy expenditure can be more than twice the normal one and repeated impact may potentially alter bone metabolism but to the best of our knowledge, there is no study that have assessed the effects of ultra-endurance running on bone tissue, particularly in males.

The main purpose of the present project is thus to quantify supraspinal central fatigue and associated changes in cortical excitability after an extreme exercise such as a mountain ultramarathon: the Ultra-Trail du Mont-blanc, by using TMS. The secondary purpose are (i) to compare neuromuscular and biological alterations induced by a mountain ultramarathon between males and females matched by age and level of performance, (ii) to evaluate, by biological urine and blood samples, the consequences of a mountain ultramarathon on kidneys and (iii) to investigate the hormonal status and bone mineral density of a group of male and female runners who take part to this type of event regularly.

ELIGIBILITY:
Inclusion Criteria:

* participating to Mont-Blanc ultramarathon
* participation in at least two ultra-endurance races like Trail

Exclusion Criteria:

* injury within 3 months before the race
* joint pathology
* contra indication for magnetic stimulation transcranial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ultramarathon runner
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
central fatigue | Immediatly after the Mont Blanc ultramarathon
  quantify supraspinal central fatigue

SECONDARY OUTCOMES:
neuromuscular and biological alterations | Immediatly after the Mont Blanc ultramarathon
  compare neuromuscular and biological alterations induced by a mountain ultramarathon between males and females matched by age and level of performance
kidney consequences | Immediatly after the Mont Blanc ultramarathon
  Evaluate, by biological urine and blood samples, the consequences of a mountain ultramarathon on kidneys
hormonal status and bone mineral density | Immediatly after the Mont Blanc ultramarathon
  investigate the hormonal status and bone mineral density of a group of male and female runners who take part to this type of event regularly

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD, Principal Investigator — CHU SAINT-ETIENNE; Guillaume MILLET, PhD, Study Chair — Université de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France